CLINICAL TRIAL: NCT05216380
Title: ActivityLink: Clinic-to-Community Physical Activity Referrals for Cardiovascular Disease Risk Reduction in Cancer Survivors.
Brief Title: Study of Clinic-delivered Physical Activity Referrals to Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jamie Faro, Assistant Professor, University of Massachusetts, Worcester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: H00021562; 1K12HL138049-01 (NIH)
Record Dates: First submitted 2022-01-05; First posted 2022-01-31 (Actual); Results first posted 2023-08-15 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Cancer; Physical Inactivity
Keywords: Cancer; Physical Activity; Cardiovascular Disease; Referrals
MeSH Terms: conditions — Neoplasms; Sedentary Behavior; Motor Activity; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ActivityLink (Experimental): ActivityLink will be a clinic implementation program delivered to clinic staff.
  Interventions: Behavioral: ActivityLink

INTERVENTIONS:
Behavioral: ActivityLink — ActivityLink is an implementation program using:
  1. Didactic and experiential training sessions for clinic staff to conduct referrals
  2. Secure electronic referral webform to refer patients using their email address and phone number
  3. Messaging sent to the patient and provider that they have been referred to a program
  4. Clinic visual cues (flyers and paper prescription pad) to reinforce referrals
  5. Motivational messaging and booster sessions from study staff to encourage referrals and troubleshoot

SUMMARY:
Background: Cancer survivors have a greater risk of cardiovascular disease (CVD) and have low physical activity levels. Physical inactivity is one modifiable risk factor for CVD, and increased physical activity has shown a cardioprotective effect on lowering CVD risk. The objective of ActivityLink is to use an electronic referral (e-referral) implementation program for clinic staff to refer survivors to an in-person and a virtual physical activity program.

Methods: Participants in this study will include clinic staff and patients. Investigators will first conduct interviews with clinic staff and patients, followed by usability testing of a referral system with staff. The study team will then beta-test two rounds of testing using Plan, Do, Study, Act (PDSA) Cycles for clinic staff to refer patients in the clinic. Quantitative data and qualitative interviews will be collected following each PDSA cycle, with refinements made based on feedback.

Outcomes: The proposed study addresses a critical need to implement physical activity referrals into routine cancer survivorship visits.

ELIGIBILITY:
Inclusion Criteria for Aim 1a:

* Medical providers who are 1) Are a current UMass Cancer Clinic patient navigator, oncologist, radiologist, or cardiologist 2) Consent to participate in the study.
* Program leaders who are 1) In charge of implementing evidence-based physical activity program for cancer patients/survivors (LIVESTRONG at the Y); 2) Consent to participate in the study.
* Patients who receive treatments at the UMass Cancer Clinics who are 1) Are at least 18 years of age; and 2) Consent to participate in the study.

Exclusion Criteria for Aim 1a:

* Medical providers who are 1) Not currently employed at UMass Memorial Health (UMH), 2) Not involved in direct treatment of care coordination of cancer patients
* Program leaders who are 1) not involved in the implementation of an evidence-based physical activity program for cancer survivors
* Patients who are 1) Unable or unwilling to provide informed consent; 2) <18 years of age.

Inclusion Criteria for Aim 1b:

* Participants for Aim 1b are eligible if they are: 1) Are a UMass Cancer Clinic patient navigator; and 2) Consent to participate in the study.

Inclusion criteria for Aim 2:

* Clinic staff who 1) Are a current UMass Cancer Clinic staff delivering care to patients 2) Consent to participate in the study.
* Program leaders who are 1) In charge of implementing evidence-based physical activity program that clinic staff refer cancer patients/survivors to (LIVESTRONG at the Y and FitCancer); 2) Consent to participate in the study.
* Patients who receive a physical activity program referral during their survivorship care planning from UMass Cancer Clinics who are 1) Are at least 18 years of age; and 2) Consent to participate in the study.

Exclusion Criteria for Aim 2:

* Clinic staff who are 1) Not currently employed at UMass, 2) Not implementing patient treatment of care coordination of cancer patients
* Program leaders who are 1) not involved in the implementation of an evidence-based physical activity program clinic staff refer cancer survivors to
* Patients who are 1) Unable or unwilling to provide informed consent; and 2) <18 years of age

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jamie M Faro, PhD, Principal Investigator — UMass Chan Medical School
Locations (1):
- University of Massachusetts Chan Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- ActivityLink: ActivityLink will be a clinic implementation program delivered to clinic staff.
  ActivityLink: ActivityLink is an implementation program using:
  1. Didactic and experiential training sessions for clinic staff to conduct referrals
  2. Secure electronic referral webform to refer patients using their email address and phone number
  3. Messaging sent to the patient and provider that they have been referred to a program
  4. Clinic visual cues (flyers and paper prescription pad) to reinforce referrals
  5. Motivational messaging and booster sessions from study staff to encourage referrals and troubleshoot
Period: Overall Study
Arm/Group | ActivityLink
Started | 69
Patient Participants | 54
Clinician Participants | 15
Completed | 69
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | ActivityLink
Number analyzed (Participants) | 54
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 60.5 (11.8)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 42
  Male | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Number of patients referred [Count of Participants; unit: Participants] | 54

OUTCOME MEASURES:

1. Primary Outcome: The Number of Patients Referred Using the Secure Webform
Description: The number of patients clinicians referred using the secure webform
Time Frame: 12 weeks from launch of referrals (baseline)
Population: This represents the total number of patients accepting referrals from their provider. There were no data on those patients who did not accept referrals, thus we can only record the number accepted.
Measure: Count of Participants; unit: Participants
Arm/Group | ActivityLink
Number analyzed (Participants) | 54
Participants | 54

2. Secondary Outcome: Proportion of Eligible Clinic Staff Who Enroll
Description: Proportion of eligible clinic staff who enrolled in the study to deliver referrals
Time Frame: 12 weeks from launch of referrals (baseline)
Population: Clinician participants
Measure: Count of Participants; unit: Participants
Arm/Group | ActivityLink
Number analyzed (Participants) | 32
Participants | 15

3. Secondary Outcome: Proportion of Referred Patients Who Enroll in Programs
Description: Proportion of referred patients who enroll in programs
Time Frame: At study completion, within 3 months of referral completion
Population: Patients who enrolled in programs
Measure: Count of Participants; unit: Participants
Arm/Group | ActivityLink
Number analyzed (Participants) | 54
Participants | 19

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | ActivityLink
All-Cause Mortality (participants affected / at risk) | 0/54
Serious Adverse Events (participants affected / at risk) | 0/54
Other Adverse Events (participants affected / at risk) | 0/54

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-22): https://cdn.clinicaltrials.gov/large-docs/80/NCT05216380/Prot_SAP_000.pdf